CLINICAL TRIAL: NCT02284854
Title: Pharmacokinetic Interaction Study Between Eslicarbazepine Acetate and Carbamazepine in Healthy Subject
Brief Title: Pharmacokinetic Interaction Study Between Eslicarbazepine Acetate and Carbamazepine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIA-2093-129
Record Dates: First submitted 2014-11-04; First posted 2014-11-06 (Estimated); Results first posted 2015-01-08 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate; Carbamazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Day 1 to Day 8 - BIA 2-093 800 mg Day 9 to Day 14 - BIA 2-093 800 mg + CBZ 200 mg Day 15 to Day 22 - BIA 2-093 800 mg + CBZ 400 mg Day 23 to Day 35 - BIA 2-093 800 mg + CBZ 400 mg twice-daily
  Interventions: Drug: BIA 2-093; Drug: Carbamazepine
- Group B (Experimental): Day 1 to Day 8 - CBZ 200 mg Day 9 to Day 14 - CBZ 400 mg Day 15 to Day 29 - CBZ 400 mg twice-daily Day 30 to Day 35 - BIA 2-093 800 mg + CBZ 400 mg twice-daily
  Interventions: Drug: BIA 2-093; Drug: Carbamazepine

INTERVENTIONS:
Drug: BIA 2-093
  Other Names: Eslicarbazepine acetate; ESL
Drug: Carbamazepine
  Other Names: CBZ

SUMMARY:
Open-label study in two parallel groups of 20 healthy subjects each. Group A assessed the effect of CBZ on ESL pharmacokinetics, and Group B assessed the effect of ESL on CBZ pharmacokinetics.

DETAILED DESCRIPTION:
Open-label study in two parallel groups of 20 healthy subjects each. Group A assessed the effect of CBZ on ESL pharmacokinetics, and Group B assessed the effect of ESL on CBZ pharmacokinetics. Each patient participated in the study for approximately 9 weeks. The clinical portion of the study was completed in approximately 3 months. Subjects received the treatments during 35 days.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18 to 45 years inclusive;
* Body mass index (BMI) between 18 and 30 kg/m2 inclusive;
* Healthy as determined by pre-study medical history, physical examination, vital signs, and 12-lead electrocardiogram (ECG); negative tests for Hepatitis B surface Antigen (HBsAg), anti-HCVAb and Human Immunodeficiency Virus (HIV)-1 and HIV-2 Ab at screening;
* Clinical laboratory test results clinically acceptable at screening and admission to each treatment period;
* Negative screen for alcohol and drugs of abuse at screening and admission to each treatment period;
* Non-smokers or ex-smokers;
* Able and willing to give written informed consent;
* If female, not of childbearing potential by reason of surgery or, if of childbearing potential, she used a double-barrier method of contraception: 1 male barrier method [male condom] plus 1 female barrier method (diaphragm, spermicide, or intrauterine device);
* If female, had a negative urine pregnancy test at screening and admission to each treatment period.

Exclusion Criteria:

* Clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders; have a clinically relevant surgical history;
* History of relevant atopy or any drug hypersensitivity (including known hypersensitivity to ESL or other carboxamide derivatives [e.g., carbamazepine, oxcarbazepine] or any of its excipients; known hypersensitivity to drugs structurally related to carbamazepine [e.g.: tricyclic antidepressants] or any of its excipients);
* Second or third-degree atrioventricular blockade not corrected with a pace-maker or any other clinically significant abnormality in the 12-lead ECG as determined by the investigator;
* History of alcoholism or drug abuse;
* Consumed more than 14 units1 of alcohol a week;
* Significant infection or known inflammatory process on screening or admission to each treatment period;
* Acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhoea, heartburn) at the time of screening or admission to each treatment period;
* Use of medicines within two weeks of admission to first period that may affect the safety or other study assessments, in the investigator's opinion;
* Had donated or received any blood or blood products within the 3 months prior to screening;
* Vegetarians, vegans or have other medical dietary restrictions;
* Could not communicate reliably with the investigator; was unlikely to co-operate with the requirements of the study;
* Unwilling or unable to give written informed consent;
* If female, was pregnant or breast-feeding;
* If female, was of childbearing potential and did not use an accepted effective contraceptive method or used hormonal contraceptives;
* Had received an investigational drug within 3 months of screening or was currently participating in another study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2009-07; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A | Group B
Started | 23 | 20
Completed | 18 | 20
Not Completed | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group B: Day 1 to Day 8 - CBZ 200 mg Day 9 to Day 14 - CBZ 400 mg Day 15 to Day 29 - CBZ 400 mg twice-daily Day 30 to Day 35 - BIA 2-093 800 mg + 400 mg twice-daily
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 23 | 20 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 20 | 43
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Cmax (BIA 2-093) - the Maximum Plasma Concentration
Description: Reference - Day 7 following once-daily oral administration of ESL 800 mg Test - Day 35 following once-daily oral administration of ESL 800 mg
Time Frame: Day 7 to 35
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group A
Number analyzed (Participants) | 18
ng/mL
  Cmax ESL (D7 ESL 800mg) | 18601 (3164)
  Cmax ESL (D35 ESL 800mg) | 14591 (1800)

2. Primary Outcome: Cmax (CBZ) - the Maximum Plasma Concentration
Description: Reference - Day 28 following twice-daily oral administration of CBZ 400 mg Test - Day 35 following twice-daily oral administration of CBZ 400 mg
Time Frame: Day 28 to 35
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group B
Number analyzed (Participants) | 20
ng/mL
  Cmax CBZ (D28 CBZ 400 mg twice-daily) | 10414 (1896)
  Cmax CBZ (D35 CBZ 400 mg twice-daily) | 9719 (2019)

3. Primary Outcome: Cmax (CBZE) - the Maximum Plasma Concentration
Description: Reference - Day 28 following twice-daily oral administration of CBZ 400 mg twice-daily Test - Day 35 following twice-daily oral administration of CBZ 400 mg twice-daily
  CBZE - carbamazepine-epoxide is the active metabolite of CBZ
Time Frame: Day 28 to 35
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group B
Number analyzed (Participants) | 20
ng/mL
  Cmax CBZE (D28 CBZ 400 mg twice-daily) | 1562 (429)
  Cmax CBZE (D35 CBZ 400 mg twice-daily) | 1560 (332)

4. Primary Outcome: AUC0-t (BIA 2-093) - Area Under the Curve to Last Measurable Concentration for BIA 2-093
Description: as for outcome 1
Time Frame: Day 7 to 35
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Group A
Number analyzed (Participants) | 18
ng*h/mL
  AUC0-t ESL (D7 ESL 800mg) | 276836 (43062)
  AUC0-t ESL (D35 ESL 800mg) | 188648 (23897)

5. Primary Outcome: AUC0-t (CBZ) - Area Under the Curve to Last Measurable Concentration for CBZ
Description: as for outcome 2
Time Frame: Day 28 to 35
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Group B
Number analyzed (Participants) | 20
ng*h/mL
  AUC0-t CBZ (D28 CBZ 400 mg twice-daily) | 104494 (16344)
  AUC0-t CBZ (D35 CBZ 400 mg twice-daily) | 94394 (17230)

6. Primary Outcome: AUC0-t (CBZE) - Area Under the Curve to Last Measurable Concentration for CBZE
Description: Reference - Day 28 following twice-daily oral administration of CBZ 400 mg Test - Day 35 following twice-daily oral administration of CBZ 400 mg
  CBZE - carbamazepine-epoxide is the active metabolite of CBZ
Time Frame: Day 28 to 35
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Group B
Number analyzed (Participants) | 20
ng*h/mL
  AUC0-t CBZE (D28 CBZ 400 mg twice-daily) | 15322 (3857)
  AUC0-t CBZE (D35 CBZ 400 mg twice-daily) | 14953 (3121)

ADVERSE EVENTS:
Groups:
- CBZ 200 mg: Group B CBZ 200 mg
- CBZ 400 mg: Group B CBZ 400 mg
- CBZ 400 mg Twice-daily: Group B CBZ 400 mg twice-daily
- ESL 800 mg + CBZ 400 mg Twice-daily: Group A + B ESL 800 mg + CBZ 400 mg twice-daily
- ESL 800 mg: Group A ESL 800 mg
- ESL 800 mg + CBZ 200 mg: Group A ESL 800 mg + CBZ 200 mg
- ESL 800 mg + CBZ 400 mg: Group A ESL 800 mg + CBZ 400 mg
- Before Treatment: Group A and B Before treatment
- After Treatment: Group A and B After treatment
Arm/Group | CBZ 200 mg | CBZ 400 mg | CBZ 400 mg Twice-daily | ESL 800 mg + CBZ 400 mg Twice-daily | ESL 800 mg | ESL 800 mg + CBZ 200 mg | ESL 800 mg + CBZ 400 mg | Before Treatment | After Treatment
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/39 | 0/23 | 0/21 | 0/19 | 0/43 | 0/38
Other Adverse Events (participants affected / at risk) | 11/20 | 9/20 | 12/20 | 21/39 | 14/23 | 10/21 | 10/19 | 0/43 | 4/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CBZ 200 mg (N=20) | CBZ 400 mg (N=20) | CBZ 400 mg Twice-daily (N=20) | ESL 800 mg + CBZ 400 mg Twice-daily (N=39) | ESL 800 mg (N=23) | ESL 800 mg + CBZ 200 mg (N=21) | ESL 800 mg + CBZ 400 mg (N=19) | Before Treatment (N=43) | After Treatment (N=38)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 2 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 3 | 2 | 0 | 2 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 3 | 4 | 7 | 5 | 7 | 3 | 0 | 0 | 0
Feeling drunk (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 2 | 1 | 0 | 1 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Inspiratory capacity abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 0 | 4 | 8 | 0 | 4 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dystonia (Nervous system disorders) | 0 | 0 | 1 | 5 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 5 | 2 | 3 | 9 | 4 | 1 | 2 | 0 | 2
Paraesthesia (Nervous system disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 4 | 1 | 5 | 5 | 4 | 0 | 0 | 0 | 0
Speech disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Menstrual discomfort (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Sweat gland disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other